CLINICAL TRIAL: NCT00827320
Title: A Single Dose, 2-Period, 2-Treatment, 2-Way Crossover Bioequivalency Study of Levetiracetam 1g Tablets Under Fed Conditions
Brief Title: Bioequivalency Study of Levetiracetam 1g Tablets Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Roxane Laboratories (Industry)
Responsible Party: Elizabeth Ernst, Roxane Laboratories, Inc.
Organization: West-Ward Pharmaceutical (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: LEVE-T1000-PVFD-1
Record Dates: First submitted 2009-01-15; First posted 2009-01-22 (Estimated); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Seizures
MeSH Terms: conditions — Seizures | interventions — Levetiracetam

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Drug: Levetiracetam — 1000 mg tablet
  Other Names: KEPPRA

SUMMARY:
The objective of this study was to prove the bioequivalence of Levetiracetam 1000 mg Tablets under fed conditions

ELIGIBILITY:
Inclusion Criteria:

* No clinically significant abnormal findings on the physical examination, medical history, or clinical laboratory results during screening

Exclusion Criteria:

* Positive test for HIV, Hepatitis B, or Hepatitis C. Treatment with known enzyme altering drugs. History of allergic or adverse response to Levetiracetam or any comparable or similar product.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 26 (Actual)
Dates: Start 2007-06; Primary Completion 2007-06 (Actual); Study Completion 2007-06 (Actual)

PRIMARY OUTCOMES:
bioequivalence based on Cmax | 10 days

CONTACTS AND LOCATIONS:
Overall Officials: Soran Hong, MD, Principal Investigator — Novum Pharmaceutical Research Services
Locations (1):
- Novum Pharmaceutical Research Services, Houston, Texas, United States